CLINICAL TRIAL: NCT03539575
Title: CB1R Availability in Synthetic Psychoactive Cannabinoid Users
Brief Title: CB1R in Synthetic Psychoactive Cannabinoids
Acronym: CB1R in Spice
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1308012514A; 1R21DA041580-01A1 (NIH)
Record Dates: First submitted 2018-03-06; First posted 2018-05-29 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Drug Dependence
Keywords: K2; Spice; Synthetic Marijuana
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Synthetic Psychoactive Cannabinoid Users (Other): Synthetic Psychoactive Cannabinoid dependent subjects who are frequent spice/K2 users will receive the radiotracer [11-C]OMAR.
  Interventions: Other: [11-C]OMAR

INTERVENTIONS:
Other: [11-C]OMAR — The radiotracer, [11-C]OMAR will be administered at no more than 10 micrograms at the beginning of each PET scan.

SUMMARY:
The purpose of this research study is to determine whether the CB1R availability is lower in synthetic psychoactive cannabinoid subjects using the most widely available synthetic psychoactive cannabinoids at the time the study is initiated.

ELIGIBILITY:
Inclusion:

* Able to provide written consent
* Age 18-55
* Current Synthetic Psychoactive Cannabinoids consumption

Exclusion:

* MRI metal exclusions and claustrophobia
* Education completed is less than 12 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Positron Emission Tomography (PET Imaging) | Change in CB1R availability from baseline throughout one test day
  CB1R availability using [11-C]OMAR PET imaging Change in CB1R availability (e.g. volume distribution).

SECONDARY OUTCOMES:
CogState Battery | Change in CB1R availability from baseline throughout one test day
  2. Changes in Cognition during withdrawal using a computerized battery Changes in cognitive functions such as attention, memory, motor functioning, and processing speed.
Electroencephalogram | Change in CB1R availability from baseline throughout one test day
  3. Changes in brain rhythms measured by Electroencephalography Changes in electroencephalographic (EEG) brain rhythms related to information processing.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, M.D., Principal Investigator — Yale University; Mohini Ranganathan, M.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No